CLINICAL TRIAL: NCT04089007
Title: Feasibility, Acceptability and Effectiveness of the SOmNI (Sleep Outcomes, Mhealth, Wearable Sensors and Nudging Intervention) Mobile Phone App for Sleep Promotion in Adolescents: SOmNI Pilot RCT
Brief Title: Feasibility, Acceptability and Effectiveness of the SOmNI Mobile Phone App for Sleep Promotion in Adolescents
Acronym: SOmNI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Robyn Stremler, Associate Professor, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: MOP-136818
Record Dates: First submitted 2018-04-05; First posted 2019-09-13 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Sleep Deprivation
MeSH Terms: conditions — Sleep Deprivation | interventions — Control Groups

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SOmNI intervention group (Experimental): Participants will receive an iPhone with the SOmNI app and will be instructed to move their bedtime earlier by 5 minutes (from their average baseline week bedtime) on each school night (Sunday to Thursday). Participants will also be given sleep hygiene information related to the embedded features of the SOmNI app. A research assistant will help the participant to enter the appropriate goal bedtime in the SOmNI app and orient them to the features of the SOmNI app. Participants will also be instructed to aim for <1 hour difference between school night and weekend bedtimes and wake times (i.e. avoid staying up late and sleeping in on weekends).
  The SOmNI application will allow the user to graphically track sleep behaviour across the four-week intervention period as recorded by the wearable sensor (e.g. bedtimes, wake times, amount of sleep achieved will all be displayed in the app).
  Interventions: Device: SOmNI app
- Control group (Active Comparator): The research assistant will advise the participant to increase the amount of nighttime sleep achieved but will not give any sleep hygiene advice or instructions for moving their bedtime earlier.
  Interventions: Other: Control group

INTERVENTIONS:
Device: SOmNI app — In addition to allowing users to track sleep behaviours across the four-week intervention period, the SOmNI app will also provide messaging via alerts and tips to outline the importance of sleep to health, suggest optimal sleep timing/duration, and suggest sleep promotion strategies. Daily review questions in the app will help the participants link changes in sleep behaviours to changes in health outcomes. As well, when goals related to sleep extension are met, the SOmNI rewards program awards points to the participant and these points can then be redeemed in $5 increments to a maximum of $40 for gift certificates.
  Arms: SOmNI intervention group
Other: Control group — The research assistant will advise the participant to increase the amount of nighttime sleep achieved but will not give any sleep hygiene advice or instructions for moving their bedtime earlier.
  Arms: Control group

SUMMARY:
This study evaluates the acceptability, feasibility, and efficacy of an intervention using wearable sensors and a mHealth application, SOmNI, to promote sleep for adolescents. The investigators hypothesize that a behavioural intervention delivered through a mobile app will be a cost-effective and accessible method of engaging adolescents in the self-management of sleep behaviours. Participants will be randomized to either the SOmNI Intervention group or the Control group. Participants receiving the SOmNI app will attempt to incrementally move their school night bedtime earlier in the evening.

DETAILED DESCRIPTION:
Over 60% of adolescents sleep less than the 9 hours of sleep recommended for 13-18 year olds. Quality of life is reduced due to the daytime consequences of chronic sleep deprivation such as sleepiness, fatigue, low mood, and inattentiveness at school. Although this sleep debt occurs in otherwise healthy adolescents, it significantly increases their risk of development of the chronic health conditions (cardiovascular disease and depression) and forms of accidental injury (motor vehicle accidents) that place the greatest demands on our health care system. Despite increased recognition of adequate sleep as a key contributor to health, there exist few effective interventions to promote sleep in adolescents. This study is designed to determine compliance, feasibility and preliminary data on health outcomes (nocturnal sleep measured objectively by actigraphy; daytime sleepiness; anxiety; depression; unintentional injuries; morning school attendance). This study will be a pilot RCT, randomizing 76 adolescents to one of two groups (i.e. 38 per group). Study arms will include a control group and intervention group (activity monitoring device with custom application). Mobile health, user-friendly low-intensity interventions with wearable sleep sensors and tailored feedback may help many adolescents to increase the amount of sleep they achieve.

ELIGIBILITY:
Inclusion Criteria:

* enrolled in high school (grades 9 to 12)
* ages 13-17 years
* report sleeping <8 hours per weeknight (Sun-Thurs)
* endorse daytime sleepiness that interferes with their daily function to a moderate or severe degree (e.g. To what extent do you consider your sleepiness to interfere with your daily functioning (e.g. daytime fatigue, mood, ability to function at school, concentration, memory)
* report sleeping >9 hours on weekend nights (Fri-Sat)
* have either their own iPhone (version 4S or higher) or are willing to use a study-provided iPhone

Exclusion Criteria:

* developmental delay (e.g. more than one grade level beyond what is appropriate for age)
* physician-diagnosed, significant physical health problem (e.g. cystic fibrosis, diabetes, lupus, kidney disease, hypertension, inflammatory bowel disease, etc)
* physician-diagnosed mental health problem (e.g. anxiety, depression, ADHD),
* physician-diagnosed sleep disorder (e.g. narcolepsy, obstructive sleep apnea, insomnia, restless leg syndrome)
* suspected sleep disordered breathing problem as identified by screening with questions from the Pediatric Sleep Questionnaire
* suspected insomnia based on screening with questions from the Insomnia Severity Index
* suspected Restless Leg Syndrome based on screening with the International RLS Study Group questionnaire
* suspected delayed sleep phase syndrome as evidenced by consistent inability to fall asleep before 01h00 to 06h00, significant impairment in the ability to attend school due to extreme delay of their sleep schedule, and avoidance of other social or family functions in the daytime

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 65 (Actual)
Dates: Start 2018-01-26 (Actual); Primary Completion 2018-06-28 (Actual); Study Completion 2018-06-28 (Actual)

PRIMARY OUTCOMES:
Compliance rate | Through study completion, an average of 6 weeks
  Compliance rate (percentage of participants assigned to intervention group who used SOMNI app to monitor sleep)
Dropout rate | Through study completion, an average of 6 weeks
  Dropout rate (percentage of participants who withdrew from the study groups)

SECONDARY OUTCOMES:
Recruitment rate | Through study completion, an average of 6 weeks
  Percent of those eligible approached to participate who gave consent
Data completion rates | Through study completion, an average of 6 weeks
  Percent of participants who completed study measurements (actigraphy, sleep diary)

OTHER OUTCOMES:
Change in nocturnal school night sleep duration | Baseline (week 1) to Follow up (week 5)
  Mean minutes of nocturnal (9pm to 9am) school night sleep (averaged over 5 nights Sun-Thurs)
Change in nocturnal weekend sleep duration | Baseline (week 1) to Follow up (week 5)
  Mean minutes of nocturnal (9pm to 9am) weekend sleep (averaged over two nights -Fri-Sat)
Change in daytime school night sleep | Baseline (week 1) to Follow up (week 5)
  Mean minutes of daytime (9am to 9pm) school night sleep (averaged over five days -Mon-Fri)
Change in daytime weekend sleep | Baseline (week 1) to Follow up (week 5)
  Mean minutes of daytime (9am to 9pm) weekend sleep (averaged over two days -Sat-Sun)
Change in daytime sleepiness | Baseline (week 1) to Follow up (week 5)
  Epworth Sleepiness Scale (minimum to maximum scores range from 0-24; values >10 represent excessive daytime sleepiness)
Change in sleep quality | Baseline (week 1) to Follow up (week 5)
  School sleep habits survey
Change in sleep hygiene | Baseline (week 1) to Follow up (week 5)
  Sleep Hygiene Index
Change in anxiety | Baseline (week 1) to Follow up (week 5)
  Speilberger State Trait Anxiety Inventory -State portion
Change in depression | Baseline (week 1) to Follow up (week 5)
  Center for Epidemiological Studies Depression scale (minimum to maximum scores range from 0-60; values >16 indicate possible clinical depression)
Change in unintentional injuries | Baseline (week 1) to Follow up (week 5)
  Questionnaire asking participants if they accidentally injured themselves (e.g. cuts, strains, falls) in the last 4 weeks
Change in morning school attendance | Baseline (week 1) to Follow up (week 5)
  Questionnaire asking participants if they arrived to school late on mornings in the last 4 weeks
Change in Body Mass Index | Baseline (week 1) to Follow up (week 5)
  Height (meters) and weight (kg) will be used to calculate BMI (kg/meters squared)
Change in Blood Pressure (mm Hg) | Baseline (week 1) to Follow up (week 5)
  Blood pressure will be taken using a manual sphygmomanometer

CONTACTS AND LOCATIONS:
Overall Officials: Robyn Stremler, RN, PhD, Principal Investigator — University of Toronto
Locations (1):
- University of Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No